CLINICAL TRIAL: NCT02106988
Title: Concurrent Chemotherapy and Radiation Therapy for Newly Diagnosed Patients With Stage I/II Nasal NK Cell Lymphoma
Brief Title: Concurrent Chemotherapy and Radiation Therapy for Newly Diagnosed Nasal NK Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0367; NCI-2014-01356 (Registry Identifier: NCI CTRP-Clinical Trials Registry)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma
Keywords: Lymphoma; NK cell lymphoma-nasal type; Radiation therapy; XRT; Dexamethasone; Decadron; Etoposide; VePesid; Ifosfamide; Ifex; Mesna; Mesnex; Carboplatin; Paraplatin
MeSH Terms: conditions — Lymphoma | interventions — Radiotherapy; Dexamethasone; Calcium Dobesilate; etoposide phosphate; Etoposide; Ifosfamide; Mesna; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemotherapy + Radiation Therapy (Experimental): Radiation therapy delivered for a total dose of 50.4 to 54 Gy over 28 to 30 treatments. Within seven days of starting radiotherapy, the first cycle of chemotherapy started and repeated every 3 weeks for a total of 3 cycles.
  DeVIC on day 1 of every cycle. Dexamethasone 40 mg by vein Days 1-3, Etoposide 67 mg/m2 by vein on Days 1-3, Ifosfamide 1 g/m2 by vein on Days 1-3, Mesna 0.4 g/m2 by vein on Days 1-3 with Ifosfamide, Mesna 0.6 g/m2 by vein over 24 hours daily on Days 1-3 via ambulatory pump, Carboplatin 200 mg/m2 by vein on Day 1. Cycles repeated every 21 days.
  Interventions: Radiation: Radiation Therapy; Drug: Dexamethasone; Drug: Etoposide phosphate; Drug: Ifosfamide; Drug: Mesna; Drug: Carboplatin

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy delivered for a total dose of 50.4 to 54 Gy 5 days a week for 28 to 30 treatments.
  Other Names: XRT
Drug: Dexamethasone — 40 mg by vein Days 1-3 in a 21 day cycle.
  Other Names: Decadron
Drug: Etoposide phosphate — 67 mg/m2 by vein on Days 1-3 of a 21 day cycle.
  Other Names: VePesid
Drug: Ifosfamide — 1 g/m2 by vein on Days 1-3 of a 21 day cycle.
  Other Names: Ifex
Drug: Mesna — 0.4 g/m2 by vein on Days 1-3 with Ifosfamide, 0.6 g/m2 by vein over 24 hours daily on Days 1-3 via ambulatory pump.
  Other Names: Mesnex
Drug: Carboplatin — 200 mg/m2 by vein on Day 1 of a 21 day cycle.
  Other Names: Paraplatin

SUMMARY:
The goal of this clinical research study is to learn if radiation therapy and chemotherapy can help control Stage 1 and/or 2 NK cell lymphoma. The safety of the radiation and chemotherapy combination will also be studied.

This is an investigational study. Radiation and chemotherapy are FDA approved and commercially available for patients with Stage 1 and/or 2 NK cell lymphoma. The combination of these therapies given at the same time is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Radiation Therapy:

You will receive radiation therapy 5 days a week for 28 to 30 treatments (up to 6 weeks). You will receive a separate consent form that will describe this treatment and its risks in more detail.

Study Visits During Radiation Therapy:

Every week during radiation therapy:

* You will have a physical exam.
* Blood (about 1 teaspoon) will be drawn for routine tests.

Chemotherapy Administration:

You will start Cycle 1 of chemotherapy during your first week of radiation. Each cycle will be 21-days long (or longer if it takes longer for your blood cell counts to recover). You will receive up to 3 cycles of chemotherapy.

On Days 1-3 of each cycle:

* You will receive dexamethasone by vein over about 15 minutes.
* You will receive etoposide by vein over 2 hours.
* You will receive ifosfamide by vein over 3 hours.
* Mesna is given to protect the bladder from side effects. You will receive mesna by vein as a non-stop infusion over 24 hours on Days 1-3 of each cycle.
* On Day 1 only, you will receive carboplatin by vein over 30 minutes.

Study Visits During Chemotherapy:

On or before Day 1, on Day 15 of Cycle 2, and on Day 15 of Cycle 3, blood (about 2 teaspoons) will be drawn for routine tests. You may also have an EKG, if the doctor thinks it is needed.

On or before Day 1 of Cycle 3:

* You will have an EKG, if the doctor thinks it is needed.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Length of Study:

You may receive radiation and up to 3 cycles of chemotherapy. You will no longer be able to receive chemotherapy if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over after the end-of-study and follow-up visits.

Follow-Up Visits:

You will also have routine follow-up visits every 3 months for the 1st year, every 4 month during the 2nd year, and every 6 months during the 3rd-5th years. After that, you will have follow up visits 1 time every year. At these visits, the following tests and procedures will be performed:

* Blood (about 2 teaspoons) will be drawn for routine tests.
* Any skin lesions that you may have that are related to the tumor will be measured and photographed.

If your doctor thinks it is needed, your MRI and PET/CT scans will be performed more or less often.

If you leave the study early:

* You will have CT, MRI, and PET/CT scans to check the status of the disease.
* Any skin lesions that you may have that are related to the tumor will be measured and photographed.
* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed stage I and II nasal NK cell lymphoma.
2. Adequate blood cell counts (i.e. ANC > 1000) at baseline, or willingness to accept supportive measures such as transfusions, filgrastim, and Epoetin.
3. Patients must have adequate liver function as indicated by: *Bilirubin </= 1.5 times the upper limit of normal (ULN), * Alanine transaminase (ALT) </= 2 times the (ULN) or aspartate transaminase (AST) </= 2 times the ULN, *These values must be obtained within two weeks before protocol entry.
4. Patients are required to have a serum creatinine </= 2.0 mg/dL. This value must be obtained within two weeks before protocol entry.
5. Left ventricular ejection fraction must be evaluated by nuclear medicine scan or echocardiography and measure >/= 50%.
6. Male patients must agree to use a barrier method of contraception or agree to abstain from heterosexual activity for the duration of the study.
7. Female patients must be willing to use two adequate barrier methods of contraception to prevent pregnancy or agree to abstain from heterosexual activity throughout the study or be post menopausal (free from menses > two years or surgically sterilized).
8. Female patients of childbearing potential must have a negative serum pregnancy test (BhCG) within 2 weeks of protocol entry.
9. Patients must have the ability to give informed consent.

Exclusion Criteria:

1. Patients with active Hepatitis B and/or Hepatitis C infection.
2. Patients with active infections requiring specific anti-infective therapy are not eligible until all signs of infections are resolved.
3. Patients known to be HIV positive.
4. Patients with pre-existing cardiovascular disease requiring ongoing treatment. This includes: a) Congestive heart failure class III/IV CHF per new york heart association (NYHA) criteria. b) Cardiomyopathy, c) Uncontrolled cardiac arrhythmia, d) Unstable angina pectoris, e) Recent MI (within 6 months).
5. Patients who are pregnant or breast-feeding.
6. Patients with psychiatric illness and/or social situations that would limit compliance with the study medication and requirements.
7. Prior radiation to the site of current primary disease, if re-treatment would lead to violation of known radiation dose tolerance limits for that site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01-16 (Actual); Primary Completion 2034-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From registration to disease progression or death due to disease, up to 5 years
  Progression defined as progressive disease or death due to disease. The evaluation of PFS will include all participants who receive radiation, regardless of whether they receive chemotherapy. Progression free survival measured from protocol entry.

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina Dabaja, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org